CLINICAL TRIAL: NCT01031641
Title: Refinement of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Via Cognitive Interviewing and Usability Testing
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910026; 10-C-N026
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Lymphomas; Leukemias; Multiple Cancers
Keywords: Patient-Reported Outcomes; Symptoms; Instrument Development; Adverse Events; Questionnaire; Patient Reported Outcomes
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

* Currently, National Cancer Institute treatment trials use clinical staff reporting to monitor adverse side effects. The clinical staff reports draw on items from the Common Terminology Criteria for Adverse Events (CTCAE).
* Several of the items in the CTCAE can be adapted for use in patient self-reporting of side effects. Researchers are interested in developing a patient-reported outcome (PRO) approach to the CTCAE.

Objectives:

* To develop questions that can be used to create a patient-reported outcome version of the CTCAE (PRO-CTCAE).
* To evaluate patient comprehension of and test the usefulness of the PRO-CTCAE questions among diverse groups of patients.

Eligibility:

* Individuals 18 years of age and older who are receiving chemotherapy or radiotherapy as cancer treatment.
* Participants must be able to speak and understand English.

Design:

* Researchers will conduct up to three rounds of interviews with patients currently receiving chemotherapy or radiation therapy treatments for cancer.
* Participants will be recruited independently from four different clinical treatment sites. At least 25 percent of patients will have an educational attainment of high school or less.
* Each patient will complete a two-part protocol, including a set of PROs that will be followed by a series of questions to evaluate patient comprehension, memory, perceived clarity, and judgment of the PROs.
* The research will be completed in approximately 1 hour, and participants will receive a small amount of compensation for their time and participation.

DETAILED DESCRIPTION:
Background:

The current approach to monitoring adverse symptom events in NCI-sponsored treatment trials is clinical staff reporting, using items from the Common Terminology Criteria for Averse Events (CTCAE). Of the 1,059 discrete items in the CTCAE, approximately 77 contain a subjective component sufficient enough to be amenable to patient self-reporting such as pain, fatigue, nausea,

and hair loss. There is general agreement that the patient, via a self-report, is the best source for reporting symptoms. Studies have shown that when compared to clinician reports, patients report earlier onset, greater severity, and longer duration of symptoms.

In September 2008, the NCI awarded a contract (N02-PC-85002-29; PI: Basch; Co-I: Hay) to support the development of an electronic-based and psychometrically robust patient-reported outcomes version of the symptom-related AEs listed in the CTCAE in an effort to improve the accuracy and precision of grading of this class of AEs. To achieve this goal, we will conduct cognitive interviews with 77 newly-developed PRO items that will subsequently be subjected to psychometric analysis, usability testing, and feasibility testing in a range of treatment settings among diverse groups of patients.

Objectives:

The overall goal of this proposed study is to evaluate patient comprehension of 77 newly developed PRO items in a range of treatment settings among diverse groups of cancer patients. The objectives are to evaluate: 1) patients understanding of the language and 2) the usability of the technology interface for collecting the PRO data of the PRO-CTCAE system.

Eligibility:

Patients will be eligible for the study if they are 1) aged 18 or older; 2) English-fluent; 3) undergoing chemotherapy and/or radiotherapy with curative or palliative intent; and 4) can provide informed consent.

Design:

We will conduct up to three rounds of cognitive interviews in 100 cancer patients at participating cancer centers including MSKCC, Dana Farber Cancer Institute, Duke and M.D. Anderson. After completion of the first round of interviews, results will be analyzed for problematic items. Revised items will be reviewed in subsequent rounds as needed. The final PRO-CTCAE items will proceed to usability testing. Usability testing will comprise three main components: 1) observation of users interacting with the web-based assessment system coupled with think aloud protocols and extensive field notes; 2) user feedback using semi-structured interviews and short surveys; and 3) web analytics including tracking for different web pages, with clickstream analysis. Usability testing will be conducted with 60 clinical research staff and 60 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Note: Patients meeting the below inclusion criteria who are registered to the study should be assigned by the individual enrolling/registering institution to one of the three Patient Groups as defined in Section 5.1.

* Age greater than or equal to18 years.
* Disease and treatment matching 1 of the 6 following cohorts:
* Cohort Breast: Breast cancer patients initiiating chemotherapy within the next 7 days or currently receiving chemotherapy.
* Cohort Lymphoma/Myeloma: Lymphoma/myeloma cancer patients initiating chemotherapy within the next 7 days or currently receiving chemotherapy.
* Cohort Prostate/Bladder: Metastatic prostate or bladder cancer patients initiating chemotherapy within the next 7 days or currently receiving chemotherapy.
* Cohort Lung: Metastatic or locally advanced lung cancer patients EITHER:
* initiating chemotherapy within the next 7 days or currently receiving chemotherapy; OR
* receiving daily radiation therapy for greater than or equal to 21 more days (concurrent chemotherapy allowed).
* Cohort Colorectal: Metastatic colorectal cancer patients initiating chemotherapy within the next 7 days or currently receiving chemotherapy.
* Cohort Head/Neck/Gastroesophageal: Head/neck/gastroesophageal cancer patients receiving daily radiation therapy for greater thanor equal to 21 more days (concurrent chemotherapy allowed).
* Cohort NCCCP: Cancer patients with cancer type NOT matching one of the previous six cohorts listed above and enrolled through an NCCCP site. Patient must be initiating active anti-cancer treatment (chemotherapy, targeted agents/biologics, and/or radiation therapy; hormonal therapy alone is not allowed) within the next 7 days or currently receiving active anti-cancer treatment (chemotherapy, targeted agents/biologics, and/or radiation therapy; hormonal therapy alone is not allowed).

NOTE: A patient registered through an NCCCP site matching one of the previous six cohorts should be registered through that cohort. Only NCCCP patients NOT matching one of the previous six cohorts should be registered through this cohort.

* Willing to return to registering institution in 1-6 weeks.
* ECOG Performance Status (PS):0-4.
* Ability to understand English and read questions on a computer screen (or listen to questions via headphones and then select responses on a screen).
* Ability to hear and respond to questions in English using a telephone keypad.

NOTE: Required for patients enrolling in Groups A and B only; not required for Group C.

* Ability to complete questionnaire(s) by themselves or with assistance.
* Provide informed written consent.
* Willing to be reached at a single telephone number (without extension or operator involvement) for the next 21 to 28 days. NOTE: Required for patients enrolling in Groups A and B only; not required for Group C.

EXCLUSION CRITERIA:

- Clinically significant cognitive or memory impairment in the opinion of clinical or research staff.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving chemotherapy or radiation treatment.@@@
Sampling Method: Probability Sample
Enrollment: 1448 (Actual)
Dates: Start 2009-11-19 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Evaluate patients understanding of measurement tool items | Study completion
  Patient report of symptom experience
Evaluate the usability of the technology interface for collecting the PRO data of the PRO-CTCAE system | Study completion
  Patient report of technology usability

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Castro, R.N., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Clark MA, Armstrong G, Bonacore L. Measuring sexual orientation and gender expression among middle-aged and older women in a cancer screening study. J Cancer Educ. 2005 Summer;20(2):108-12. doi: 10.1207/s15430154jce2002_12. PMID 16083375
- [Background] Diefenbach MA, Weinstein ND, O'Reilly J. Scales for assessing perceptions of health hazard susceptibility. Health Educ Res. 1993 Jun;8(2):181-92. doi: 10.1093/her/8.2.181. PMID 10148827
- [Background] Friedenreich CM, Courneya KS, Bryant HE. Relation between intensity of physical activity and breast cancer risk reduction. Med Sci Sports Exerc. 2001 Sep;33(9):1538-45. doi: 10.1097/00005768-200109000-00018. PMID 11528344
- [Derived] Atkinson TM, Reeve BB, Dueck AC, Bennett AV, Mendoza TR, Rogak LJ, Basch E, Li Y. Application of a Bayesian graded response model to characterize areas of disagreement between clinician and patient grading of symptomatic adverse events. J Patient Rep Outcomes. 2018 Dec 4;2(1):56. doi: 10.1186/s41687-018-0086-x. PMID 30515599
- [Derived] Schoen MW, Basch E, Hudson LL, Chung AE, Mendoza TR, Mitchell SA, St Germain D, Baumgartner P, Sit L, Rogak LJ, Shouery M, Shalley E, Reeve BB, Fawzy MR, Bhavsar NA, Cleeland C, Schrag D, Dueck AC, Abernethy AP. Software for Administering the National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events: Usability Study. JMIR Hum Factors. 2018 Jul 16;5(3):e10070. doi: 10.2196/10070. PMID 30012546